CLINICAL TRIAL: NCT00160394
Title: Multi-Centre, Single-Blind, Parallel Group, Clinical Evaluation of the Efficacy and Safety of Duac® Gel And Differin® Gel in the Topical Treatment of Mild to Moderate Acne Vulgaris
Brief Title: Comparison of Duac® Gel And Differin® Gel in Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S194-INT-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
Keywords: Mild to Moderate
MeSH Terms: conditions — Acne Vulgaris

INTERVENTIONS:
Drug: Duac® Gel / Differin® Gel

SUMMARY:
Comparing the efficacy and safety of a gel formulation containing a combination of clindamycin phosphate (equivalent to 1% clindamycin) and benzoyl peroxide (5%) once daily with a gel containing 0.1% adapalene once daily in the treatment of acne vulgaris of mild to moderate severity.

DETAILED DESCRIPTION:
Title: A Multi-Centre, Single-Blind, Parallel Group, Clinical Evaluation of the Efficacy and Safety of Duac® Gel (a Gel Containing Clindamycin Phosphate [Equivalent to 1% Clindamycin] and 5% Benzoyl Peroxide) And Differin® Gel (a Gel Containing 0.1% Adapalene) in the Topical Treatment of Mild to Moderate Acne Vulgaris

Objectives: To compare the efficacy and safety of a gel formulation containing a combination of clindamycin phosphate (equivalent to 1% clindamycin) and benzoyl peroxide (5%) once daily with a gel containing 0.1% adapalene once daily in the treatment of acne vulgaris of mild to moderate severity.

Study methodology: Randomised, comparator-controlled, single-blind trial. The Investigators/ Assessors will be blinded to the treatment received.

Study population: Male and female patients, aged 12-39, with mild to moderate acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild to moderate acne vulgaris of the face with at least 15 inflammatory lesions and/or non-inflammatory lesions, but no more than three nodulocystic lesions and an acne grade of greater than 2.0 and less than 7.0 (The Leeds Revised Acne Grading System7).
2. Patients of either sex aged between 12 and 39 years, inclusive.
3. Patients who are willing and able to provide written informed consent, after being informed of all the pertinent aspects of the trial. In the case of patients aged under 16 years of age, parental or guardian consent must be obtained in addition to patient assent.
4. Patients agreeing not to use sun-beds or undergo any UV light treatment for 4 weeks prior to entering the study and to minimise the amount of exposure to direct sunlight for the duration of the study.
5. Patients agreeing to minimise their alcohol consumption throughout the study, with a limit of 14 units per week.

Exclusion Criteria:

1. Female patients who are pregnant, breast-feeding, or sexually active and not using reliable contraception and/or not prepared to do so for the duration of the trial (a negative pregnancy test must be confirmed at Visit 1 and at the end of the study, for all females if menarche has occurred).
2. Patients using anti-androgen containing contraceptives.
3. Patients who, during the past month, have received oral or topical steroids, oral or topical antibiotics, or acne treatment of any type, including natural or artificial UV therapy.
4. Patients who have a history of hypersensitivity or idiosyncratic reaction to clindamycin phosphate, benzoyl peroxide, adapalene or any components of the study medications.
5. Patients using, or having used in the past month, any significant concomitant medication which might affect their acne, as judged by the Investigator.
6. Patients with severe systemic diseases (e.g., severely impaired renal or liver function, severe cardiovascular, neurological disease, or any other diseases that may interfere with the evaluation of the study medications). This also applies to patients with psoriasis, acne rosacea, allergic rashes, bacterial, viral or fungal infections of the facial skin, or other diseases of the facial skin.
7. Patients with a history of regional enteritis or ulcerative colitis, or a history of antibiotic-associated colitis.
8. Patients who have a history of photosensitivity.
9. Patients who are unreliable or unlikely to be available for the duration of the follow-up.
10. Patients who have participated in a clinical trial involving a drug within 30 days of recruitment into the study (or are likely to do so at any time during their participation).
11. Patients who are either an immediate family member, or a colleague, of study personnel.
12. Patients who already have a member of their household entered onto this trial.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2004-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline of inflammatory lesion counts at week 2

SECONDARY OUTCOMES:
Absolute change from baseline of inflammatory lesion counts at week 2.
Absolute change and percentage change from baseline of inflammatory lesion counts at weeks 1, 4, 8 and 12.
Absolute change and percentage change from baseline of non-inflammatory lesion counts and total lesion counts at weeks 1, 2, 4, 8 and 12.
Also, acne grade and global change score at weeks 1, 2, 4, 8 and 12 will be investigated.
Patient's self-rating assessment at weeks 1, 2, 4, 8 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: A Chu, MB BS, FRCP, Principal Investigator — Hammersmith Hospital, London; A Langner, MD, DSc, Principal Investigator — Iwolang spoo, Warsaw
Locations (3):
- Prof A Langner, Warsaw, Poland
- United Kingdom (2):
  - Dr V Goulden, Leeds
  - Dr A Chu, London